CLINICAL TRIAL: NCT06532227
Title: AspergillusOne-Health: Deciphering Azole Resistance in Aspergillus Fungi Using a One Health Approach
Acronym: AspergillusOH
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0008
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Aspergillus Fumigatus Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group control : patient without resistance: control patients with susceptible Aspergillus.
  Interventions: Other: No intervention
- Group resistant : patient without resistance: Cases are patients with resistant Aspergillus
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention excepted data collection

SUMMARY:
During a two year prospective study onpatients from department's hospitals and centralized by the pneumology department Nantes CH,all respiratory clinical samples will be cultivated for Aspergillus isolation (2900Aspergillusisolates) as standard care. The azole susceptibility pattern of isolates will be determined to itraconazole, voriconazole by subculture on azole- enriched medium at 35°c as primary screen and resistance confirmed by EUCAST Reference metho.In parallel, the relevance of detecting resistance (TR34 and TR46) directly in culture-negative BAL respiratory samples by a qPCR method will be studied in an attempt to reach a greater exhaustiveness of the resistance phenomeno. In case of azole-resistant isolate,patient data such as the underlying disease,date and site of Aspergillus isolation,disease classification,previous azole drug exposure,and home and work geographic allocation,occupation of the patient will be collecte. For all other aspergillus occurrences, underlying disease, previous azole drug exposure,home and work location of the patient will be collected in an attempt to identify risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient who has given his or her consent to participate in the study
* Patient affiliated to a social security scheme
* Patient with a respiratory sample taken between 2020 and 2023 for the retrospective cohort and from 2024 for the prospective cohort in which Aspergillus has been isolated
* Patients living in the Loire Atlantique and Vendée regions

Exclusion Criteria:

* Patient under guardianship or legal protection
* Patient of no fixed adress

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective inclusion of patients sampled as part of their care in a pneumology department (Nantes University Hospital or CHD Vendée) who are carriers of aspergillus. Patients will be contacted by email or paper mail if a strain is isolated.
  Only patients with resistant strains and susceptible patients matched to resistant strains for this study will also receive a home visit from the CMEI (except for patients living in institutions).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Environmental risk factors | 24 months
  Identify the "macro" environmental risk factors for acquiring azole-resistant aspergillus.

SECONDARY OUTCOMES:
Describe the management and evolution of resistant | 48 months
  Clinical information from each additional patient visit and presence or absence of resistant Aspergillus in home samples.
Risk factors | 48 months
  Identify individual risk factors linked to the immediate environment in the patient's home, drug management, between cases and matched controls, etc..